CLINICAL TRIAL: NCT03621995
Title: Oxidative Stress in Testicular Tissue Before and After Cryopreservation
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya Hasan, Resident in dermatology department, Assiut University
Other Study IDs: OSITTBAAC
Record Dates: First submitted 2018-07-20; First posted 2018-08-09 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Oxidative Stress
MeSH Terms: interventions — Malondialdehyde

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

GROUPS / COHORTS (3):
- Obstructive azoospermia: Malondialdehyde and Catalase level measurement before and after cryopreservation
  Interventions: Other: Malondialdehyde and Catalase level measurement
- Non obstructive azoospermia: Malondialdehyde and Catalase level measurement before and after cryopreservation
  Interventions: Other: Malondialdehyde and Catalase level measurement
- Negative group: Malondialdehyde and Catalase level measurement without cryopreservation
  Interventions: Other: Malondialdehyde and Catalase level measurement

INTERVENTIONS:
Other: Malondialdehyde and Catalase level measurement — Malondialdehyde and Catalase level measurement by colorimetric method

SUMMARY:
The absence of sperms in ejaculated semen, is the most severe form of male-factor infertility and is present in approximately 5 % of all investigated infertile couples.

DETAILED DESCRIPTION:
Obstructive azoospermia is defined as the absence of spermatozoa in the ejaculate despite normal spermatogenesis.Infection, Iatrogenic injury, Vasectomy and congenital atresia are the possible causes of it. Non obstructive or functional azoospermia results from testicular failure, which is the absence or inadequate production of fully developed spermatozoa within the testes.

Etiologies for testicular failure include genetic disorders such as sexual chromosomal abnormalities ; translocations and microdeletions of the Y chromosome; cryptorchidism; testicular torsion; radiation and toxins.

The advent of intra-cytoplasmic sperm injection has transformed the treatment of this type of severe male-factor infertility.

Surgical techniques for sperm retrieval:Testicular sperm aspiration: In men with obstructive azoospermia ,testicular sperm aspiration invariably generates enough sperm for intra-cytoplasmic sperm injection.

Testicular sperm extraction:This conventional method of surgical sperm extraction generally offers the best chance of retrieving spermatozoa, especially in functional cases and when guided by surgical microscope. However, it can be done by simple open conventional biopsy and closed surgical extraction resembling Trucut biopsy using a special cannula.

Cryopreservation Cryopreservation of human testicular tissue obtained by biopsy can be used as a potential future source of sperms. For adult cancer survivors, cryopreservation of testis biopsies may be the only option remaining if they prefer to father their own biological progeny.

There are 4 types of cryopreservation :

Slow freezing: involves step-wise programmed decrease in temperature. Rapid freezing: was first proposed by . Ultra-rapid freezing :can be considered midway technique between slow freezing and vitrification.

Vitrification: solidifies the sample into a glass-like state. During the freezing process,increasing in susceptibility of spermatozoa to lipid peroxidation,as affected by cold shock, plays an important role in ageing of spermatozoa ,shortening their lifespan and affecting the preservation of semen.The major susceptibility is related in, part to the content of polyunsaturated fatty acids.

Oxidative stress and antioxidants: Oxygen is required to support life, but its metabolites, such as reactive oxygen species, can modify cell functions and endanger cell survival. For this reason,reactive oxygen species is inactivated continuously to maintain only the small amount necessary to maintain normal cell function. There is a balance between the different antioxidants and oxidants at normal status. Oxidative stress is a cellular condition associated with an imbalance between the production of free radicals, mainly reactive oxygen species, and the scavenging capacity of antioxidants.

Superoxide dismutase and catalase are endogenous antioxidants, which protect cells from oxidative stress. Scavengers of reactive oxygen species and antioxidants are important in treating and preventing the damage caused by such stress.

Catalase has been reported from testis, seminal plasma, and spermatozoa Tissue level of malondialdehyde is proven indicator of oxidative stress resulting from lipid peroxidation .

The process of cryopreservation is known to cause more production and/or accumulation of reactive oxygen species, as antioxidant defenses are reduced in the process.

ELIGIBILITY:
Inclusion Criteria:

- Men with azoospermia at reproductive age .

Exclusion Criteria:

* Pyospermia.
* Previous trial of cryopreservation.
* Systemic diseases.
* Cryptorchidism history.
* Smoking

Ages: 14 Years to 80 Years | Sex: Male
Age Groups: Child, Adult, Older Adult
Study Population: 45 patients complaining of azoospermia who attended to the Andrology Outpatient Clinic, Dermatology ,Venerology and Andrology department, Assuit University Hospital, Assuit ,Egypt .Patients were divided into 3 groups:
  * Group A : 15 patients with obustructive azoospermia and positive testicular samples for sperms .
  * Group B : 15 patients with non obustructive azoospermia and positive testicular samples for sperms.
  * Group C : 15 patients with azoospermia and negative testicular samples for spems.
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Measurement of the level of oxidative stress that is caused by cryopreservation of testicular tissue. | 3 years
  Evaluation of oxidative stress caused by cryopreservation of testicular tissue by measurement of :
  1. Catalase activity as one indicator of antioxidants by colorimetric method.
  2. Malondialdehyde level as one indicator of lipid peroxidation by colorimetric method.

CONTACTS AND LOCATIONS:
Overall Officials: Aya H Younis, Resident, Principal Investigator — Assiut University
Locations (1):
- Assuit University Hospital, Asyut, Egypt